CLINICAL TRIAL: NCT02642094
Title: Aging Mammary Stem Cells and Breast Cancer Prevention
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early according to the protocol due to efficacy.
Sponsor: LuZhe Sun (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, LuZhe Sun, Co-Principal Investigator, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CTMS 15-2096; 1R01CA192564-01A1 (NIH)
Record Dates: First submitted 2015-11-25; First posted 2015-12-30 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Cancer of Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- The effect of short-term rapamycin treatment (Experimental): Subjects will be given a low dose of rapamycin at 2 mg/day for 5-7 days of treatment. A surgical specimen will be taken 3-7 days after the last dose of rapamycin. The specimens will be evaluated for lesion size, nuclear grade, presence of necrosis in each patient's core biopsy and surgical specimens, as well as IHC (ImmunoHistoChemistry) for biomarkers including p16, COX2 (cyclooxygenase-2), and Ki-67. Specimens will also be tested for rapamycin treatment on the properties of mammary stem/progenitor cells as another biomarker for gauging the efficacy of rapamycin treatment.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Low dose of rapamycin at 2 mg/day for -5-7 days of treatment
  Other Names: Sirolimus

SUMMARY:
To examine whether rapamycin can reduce malignant markers and aberrant mammary stem/progenitor cells (MaSCs) number in surgical specimens

DETAILED DESCRIPTION:
A non-randomized, open-label, phase II, window of opportunity trial will be carried out to see if a 5-7 day rapamycin treatment can reduce malignant markers and aberrant MaSC number

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed menopausal status. All patients who have NOT had a prior bilateral oophorectomy and/or are younger than age 60, will require menopausal status verified by FSH and estradiol local labs.
* Women diagnosed with DCIS/LCIS, Atypical lobular hyperplasia (ALH) or ADH lesions detected by pathology
* Women scheduled for mastectomy or lumpectomy after DCIS/LCIS, ALH or ADH diagnosis
* Women consented to the UT Health Cancer Center MD Anderson Cancer Center tissue biorepository (HSC20070684H)
* Women of child-bearing potential willing to practice 2 forms of contraception, one of which must be a barrier method until at least 30 days after the last dose of rapamycin.
* Women of child-bearing potential must have a negative serum pregnancy test at time of enrollment.
* Patients must be able to swallow and retain oral medication.
* All patients must have given signed informed consent prior to registration on study.
* Patients must have normal organ and marrow function as defined below:

  1. Leukocytes ≥ 3,000/uL
  2. Absolute neutrophil count ≥ 1,500/uL
  3. Platelets ≥ 100,000/uL
  4. AST ≤ 2.5 X ULN
  5. ALT ≤ 2.5 X ULN
  6. Total bili ≤ 1.5 X ULN or Direct bili ≤ 1 X ULN

Exclusion Criteria:

* Women who are pregnant.
* Women who are receiving any other concomitant treatment for their DCIS/LCIS, ALH or ADH
* Women who are taking rapamycin for another diagnosis.
* Women with an allergy to rapamycin or its derivatives.
* Active infection requiring systemic therapy.
* Patients who are taking any pills containing herbal (alternative) medicines are NOT eligible for participation. Patients must be off any such medications by the time of registration.
* Immunocompromised subjects, including patients with human immunodeficiency virus
* Women currently taking strong CYP3A4 inducers or inhibitors. Drugs that cannot be coadministered with rapamycin include but are not limited to: Calcium channel blockers: nicardipine, Antifungal agents: clotrimazole, fluconazole, Antibiotics: troleandomycin, Gastrointestinal prokinetic agents: cisapride, metoclopramide, Other drugs: bromocriptine, cimetidine, danazol, HIV-protease inhibitors (e.g., ritonavir, indinavir), Anticonvulsants: carbamazepine, phenobarbital, phenytoin, Antibiotics: rifapentine. The research team can provide a full list of these medications.
* Patients with any of the following conditions or complications are NOT eligible for participation:

  1. GI tract disease resulting in an inability to take oral medication
  2. Malabsorption syndrome
  3. Require IV alimentation
  4. History of prior surgical procedures affecting absorption
  5. Uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LuZhe Sun, PhD, Principal Investigator — University of Texas Health Science Center San Antonio, Co-PI; Ismail Jatoi, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Bouamar H, Broome LE, Lathrop KI, Jatoi I, Brenner AJ, Nazarullah A, Gorena KM, Garcia M, Chen Y, Kaklamani V, Sun LZ. mTOR inhibition abrogates human mammary stem cells and early breast cancer progression markers. Breast Cancer Res. 2023 Oct 30;25(1):131. doi: 10.1186/s13058-023-01727-z. PMID 37904250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We acquired primary tissue samples from patients diagnosed with non-invasive lesions as detected by clinical pathology at the University of Texas Health Science Center at San Antonio (UTHSCSA) (San Antonio, TX). Inclusion criteria and exclusion criteria were descried in the study.
Groups:
- Rapamycin Treatment Group: Patients with stage zero breast cancer were given a low dose of rapamycin at 2 mg/day for 5-7 days of treatment. A surgical specimen will be taken 3-7 days after the last dose of rapamycin. The specimens were evaluated with IHC (ImmunoHistoChemistry) for cancer progression biomarkers including p16, COX2 (cyclooxygenase-2), and Ki-67. Specimens were tested for rapamycin treatment on the properties of mammary stem/progenitor cells as another biomarker for gauging the efficacy of rapamycin treatment.
  A total of 40 patients were consented to undergo treatment and 38 successfully completed the regiment. The control group included 12 patients with DCIS or ADH, who declined to participate in the sirolimus study but agreed to donate their tissues, and 6 patients with invasive ductal carcinoma for a total of 18 controls.
  Rapamycin: Low dose of rapamycin at 2 mg/day for -5-7 days of treatment
- Un-treated Control Group: Subjects that consented to provide tissue, but were not treated with Rapamycin
Period: Overall Study
Arm/Group | Rapamycin Treatment Group | Un-treated Control Group
Started | 40 | 18
Completed | 38 (We enrolled 40 patients as of Feb. 2022, which is 67% of planned enrollment. Since COVID-19 started, it had been very difficult to enroll patients and to keep them on schedule for surgery, which was considered non-essential surgery and was often postponed.) | 18
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: This was a non-random, open-label, phase II, window of opportunity trial to investigate a possible inhibition of mammary stem cells (MaSCs) in non-cancerous tissue and/or malignant markers by rapamycin in patients with non-invasive breast cancer. A total of 40 patients agreed to undergo the treatment and 38 successfully completed the regiment. The control group for providing non-cancerous breast tissue included 12 patients with non-invasive breast cancer and 6 with invasive cancer.
Groups:
- Rapamycin Treatment Group: A total of 40 patients were consented to undergo treatment and 38 successfully completed the regiment.
- Un-treated Control Group: The control group included 12 patients with DCIS or ADH, who declined to participate in the sirolimus study but agreed to donate their tissues, and 6 patients with invasive ductal carcinoma for a total of 18 controls
- Total: Total of all reporting groups
Arm/Group | Rapamycin Treatment Group | Un-treated Control Group | Total
Number analyzed (Participants) | 40 | 18 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 3 | 32
  >=65 years | 11 | 15 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 18 | 58
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 9 | 33
  Not Hispanic or Latino | 14 | 8 | 22
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 33 | 15 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 40 | 18 | 58

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Short-term Rapamycin Treatment on Biomarker Ki67 Associated With Progression to Invasive Breast Cancer
Description: Comparing biopsy tissues before the treatment with surgical samples after rapamycin treatment in the same individuals to determine percentage nuclei with positive staining for Ki67 in the CCIS lesions.
Time Frame: Baseline to 5-7 day rapamycin plus 3-7 day washout
Population: Tissue samples were randomly selected from 12 patients with DCIS who participated in the treatment study
Measure: Mean (Standard Deviation); unit: percentage of Ki67+ cells
Groups:
- Effect of Short-term Rapamycin Treatment on Biomarker Ki67: Biopsy samples from patients diagnosed with DCIS to determine the effect of short-term rapamycin treatment on biomarker Ki67
Arm/Group | Effect of Short-term Rapamycin Treatment on Biomarker Ki67
Number analyzed (Participants) | 12
percentage of Ki67+ cells
  Pre-treatment | 8.235 (5.848)
  Post-treatment | 3.666 (3.176)
Statistical Analysis 1: Comparison: Effect of Short-term Rapamycin Treatment on Biomarker Ki67; Test type: Superiority; p = 0.0020, t-test, 2 sided

2. Primary Outcome: The Effect of Short-term Rapamycin Treatment on the Frequency of Luminal Progenitor Epithelial Cells
Description: Assessment will be used to measure changes in luminal progenitor cell population between controls and treated patients.
Time Frame: 5-7 day rapamycin treatment plus 3-7 day washout for the treatment group.
Population: We were only able to obtain fresh surgical tissues and mammary epithelial cell profiles by flowcytometry from 27 patients in the treatment group. The mean data of luminal progenitor cells were compared between the control and treatment groups with unpaired t test.
Measure: Mean (Standard Deviation); unit: percentage of total lineage neg. cells
Groups:
- Control: Adjacent breast tissues from control group were used for measuring the frequency of basal, luminal progenitor, and mature luminal epithelial cells.
- Treatment Group: Adjacent breast tissues from the treatment group were tested for the effect of rapamycin treatment on the frequency of basal, luminal progenitor, and mature luminal epithelial cells.
Arm/Group | Control | Treatment Group
Number analyzed (Participants) | 18 | 27
percentage of total lineage neg. cells | 11.82 (9.221) | 6.178 (5.525)
Statistical Analysis 1: Comparison: Control vs Treatment Group; Test type: Superiority; p = 0.0137, t-test, 2 sided

3. Primary Outcome: The Effect of Short-term Rapamycin Treatment on Sphere Formation Efficiency of Mammary Stem Cells
Description: Measurement of difference in sphere formation efficiency (SFE) by mammary stem cells (MaSCs) in the basal myoepithelial cell population between the control and treatment groups. SFE is an in vitro method by quantifying the number of spheres formed divided by the number of cells seeded. Higher SFE indicates higher frequency of MaSCs.
Time Frame: 5-7 day rapamycin treatment plus 3-7 day washout for the treatment group.
Population: We were only able to obtain fresh surgical tissues and mammary epithelial cell profiles by flowcytometry from 27 patients in the treatment group. Out of the 27, only 22 samples yielded enough basal myoepithelial cells for the quantification of the SFE. Comparison between control group and treatment group.
Measure: Mean (Standard Deviation); unit: spheres formed per 1,000 cells
Groups:
- Control: Adjacent breast tissues from control group were used for measuring the MaSC frequency in basal myoepithelial cells.
- Treatment Group: Adjacent breast tissues from the treatment group were used for measuring the MaSC frequency in basal myoepithelial cells.
Arm/Group | Control | Treatment Group
Number analyzed (Participants) | 18 | 22
spheres formed per 1,000 cells | 3.681 (2.303) | 0.717 (1.414)
Statistical Analysis 1: Comparison: Control vs Treatment Group; Test type: Superiority; p < 0.0001, t-test, 2 sided

4. Primary Outcome: The Effect of Short-term Rapamycin Treatment on the Frequency of Mature Luminal Epithelial Cells
Description: Measurement of Mature luminal cell populations in the treatment group compared to the control group.
Time Frame: 5-7 day rapamycin treatment plus 3-7 day washout for the treatment group.
Population: We were only able to obtain fresh surgical tissues and mammary epithelial cell profiles by flowcytometry from 27 patients in the treatment group.
Measure: Mean (Standard Deviation); unit: percentage of total lineage neg. cells
Arm/Group | Control | Treatment Group
Number analyzed (Participants) | 18 | 27
percentage of total lineage neg. cells | 11.82 (9.221) | 6.178 (5.525)
Statistical Analysis 1: Comparison: Control vs Treatment Group; Test type: Superiority; p = 0.0072, t-test, 2 sided

5. Primary Outcome: The Effect of Short-term Rapamycin Treatment on Sphere Formation Efficiency of Luminal Progenitor Cells
Description: The measurement of sphere formation efficiency (SFE) between luminal progenitor (LP) cells from the control group and those from the treatment group. SFE is an in vitro method by quantifying the number of spheres formed divided by the number of cells seeded. Higher SFE indicates higher frequency of LP cells.
Time Frame: 5-7 day rapamycin treatment plus 3-7 day washout for the treatment group.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Spheres formed from 1,000 cells
Groups:
- Control: Adjacent breast tissues from control group were used for measuring the sphere formation efficiency of luminal progenitor cells.
- Treatment Group: Adjacent breast tissues from the treatment group were used for measuring the sphere formation efficiency of luminal progenitor cells.
Arm/Group | Control | Treatment Group
Number analyzed (Participants) | 18 | 22
Spheres formed from 1,000 cells | 20.82 (20.97) | 30.32 (34.15)
Statistical Analysis 1: Comparison: Control vs Treatment Group; Test type: Superiority; p = 0.3093, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month
Description: It was used at a low dose and short term. Control group participants were not treated and therefore were not assessed for adverse events.
Groups:
- Rapamycin Treatment: Adverse events are only reported for the treatment group who received the intervention.
Arm/Group | Rapamycin Treatment
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 24/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rapamycin Treatment (N=40)
Diarrhea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 3
Headache (General disorders) | 9
Nausea (General disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Stomach pain (Gastrointestinal disorders) | 3

LIMITATIONS AND CAVEATS:
Our hypothesis was that a low dose and short term treatment with rapamycin in patients with early stage breast cancer would show significantly attenuation of mammary stem and progenitor cell activity and tumor progression biomarkers in a non-randomized study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT02642094/Prot_SAP_000.pdf